CLINICAL TRIAL: NCT00156533
Title: Long Term Treatment With Zolpidem: The Relative Efficacy of Nightly (Quaque Hora Somni [QHS]) & Intermittent Dosing and the Potential for Long Term Clinical Gains After Treatment Discontinuation.
Brief Title: Long Term Treatment With Zolpidem: Nightly and Intermittent Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Principal Investigator, Wilfred Pigeon, PhD, Assistant Professor of Psychiatry, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI Initiated; 11045 (Other: University of Rochester)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Insomnia; Primary Insomnia; Psychophysiologic Insomnia
Keywords: Insomnia; Sleep; zolpidem; Ambien; Hypnotics
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): QHS dosing with placebo (i.e. nightly dose)
  Interventions: Drug: Sugar Pill
- QHS Zolpidem (Active Comparator): QHS dosing with 10mg of zolpidem (i.e. nightly dose)
  Interventions: Drug: Zolpidem
- Intermittant Zolpidem (Experimental): Intermittent dosing with 10mg of zolpidem (3-5 pills per week as needed
  Interventions: Drug: Zolpidem
- Control (No Intervention): Monitor only condition (no placebo, no drug).

INTERVENTIONS:
Drug: Zolpidem — 10 mg of Zolpidem
  Other Names: Ambien
  Arms: Intermittant Zolpidem; QHS Zolpidem
Drug: Sugar Pill
  Arms: Placebo

SUMMARY:
We want to assess whether "how and when" one takes sleep medication results in similar or different outcomes with respect to symptom relief. We also want to know whether taking medication for a period of time provides continued benefit once the medication is stopped.

DETAILED DESCRIPTION:
To date, the aggressive treatment (Tx) of chronic insomnia has been evaluated in terms of whether maintenance therapy is possible. While what constitutes maintenance therapy is a matter of debate, there are two studies which show that benzodiazepine receptor agonists (BZRAs) 1) are effective when used intermittently for up to 3 months and 2) may be used on a nightly basis for up to 6 months with no loss of efficacy.

The significance of the present research is two fold. First, it will allow us to compare the two primary strategies used for long term treat of insomnia (nightly dosing vs intermittent dosing). Second, it will allow an evaluation of the possibility that extended treatment, given careful withdrawal from medication, may yield long term clinical gains.

Re: Objective 1: It is widely assumed that intermittent dosing confers increased efficacy. That is, less frequent medication use will extend the duration of time for which the medication is maximally potent. An empirical assessment of this proposition is required. If incorrect, physicians and patients should be encouraged to adopt a more aggressive approach to treatment. If correct, physicians and patients should be encouraged to adopt the intermittent dosing approach to treatment.

Re: Objective 2: It is widely assumed that treatment with sedatives (sleep promoting medications) constitutes only palliative care. An empirical assessment of this proposition is required. If correct, physicians and patients should be encouraged to adopt a more aggressive approach to long term treatment. If incorrect, physicians and patients should be encouraged to adopt an approach to treatment that is not currently a standard of practice: extended treatment with a clear plan to taper medication that is designed to maintain the clinical gains that occurred with medication use.

We propose to evaluate the above issues in a pilot study of 40 subjects with Primary Insomnia where subjects are randomized to one of 4 conditions:

1. QHS dosing with placebo
2. QHS dosing with 10mg of zolpidem
3. Intermittent dosing with 10mg of zolpidem (3-5 pills per week as needed)
4. Monitor only condition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25 - 55
* a stable sleep/wake schedule with a preferred sleep phase between 10:00 p.m. and 8:00 a.m.
* Patients with Primary Insomnia will meet diagnostic criteria for Psychophysiologic Insomnia according to the International Classification of Sleep Disorders manual (ICSD).
* complaint of disturbed sleep must have the following characteristics: >30 minutes to fall asleep, and/or >30 minutes wake after sleep onset time, a total sleep time of no more than 6.5 hours (or a sleep efficiency of less than 85%), a problem frequency of >4 nights/ week and a problem duration >6 months.

Exclusion Criteria:

* Unstable medical or psychiatric illness
* Use of medication that may cause insomnia or may be reduce the effectiveness of zolpidem (e.g. selective serotonin reuptake inhibitors(SSRI's), steroids, bronchodilators, calcium channel blockers, beta blockers, etc.)
* symptoms suggestive of sleep disorders other than insomnia
* polysomnographic data indicating sleep disorders other than insomnia
* Evidence of active illicit substance use or fitting criteria for alcohol abuse or dependence
* inadequate language comprehension
* pregnancy
* first-degree relatives with bipolar disorder or schizophrenia

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Perlis, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Sleep Research Laboratory, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from television and newspaper ads. After a telephone or web based screening, subjects brought into the lab to read the Informed Consent Form (ICF). After the ICF has been signed, an initial medical and psychiatric evaluation completed. If the subjects remain eligible they are required to keep two weeks of sleep diaries.
Groups:
- Placebo: Once nightly dosing (quaque hora somni [QHS])with placebo
- QHS (Nightly) Zolpidem: Once nightly (QHS) dosing with 10mg of zolpidem
- CTRL: Monitor only condition.
Period: Overall Study
Arm/Group | Placebo | QHS (Nightly) Zolpidem | Intermittant Zolpidem | CTRL
Started | 5 | 5 | 5 | 5
Completed | 3 | 3 | 3 | 3
Not Completed | 2 | 2 | 2 | 2
Not completed — Withdrawn - Medication Expiration | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Failed Screening | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: QHS dosing with placebo
- QHS Zolpidem: QHS dosing with 10mg of zolpidem
- Total: Total of all reporting groups
Arm/Group | Placebo | QHS Zolpidem | Intermittant Zolpidem | CTRL | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 5 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 4 | 14
  Male | 1 | 2 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency (SL)
Description: Number of subjects with any reduction in SL (time to fall asleep in minutes)at post-tx compared to baseline where mean SL = mean of daily values for one week calculated from sleep diary values.
Time Frame: Baseline and Post-treatment (12wks)
Population: Completers Only
Measure: Number; unit: participants
Groups:
- Placebo: QHS (i.e., nightly) dosing with placebo
- QHS Zolpidem: QHS (i.e., nightly) dosing with 10mg of zolpidem
- Intermittant Zolpidem: Intermittent dosing with 10mg of zolpidem (3-5 pills per week as needed)
- CTRL: Monitor only condition (no placebo and no zolpidem).
Arm/Group | Placebo | QHS Zolpidem | Intermittant Zolpidem | CTRL
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 1 | 2 | 3 | 0

2. Secondary Outcome: Wake After Sleep Onset (WASO)
Description: Number of subjects with any reduction in WASO at post-tx compared to baseline where mean WASO = mean of daily values for one week calculated from sleep diary values.
Time Frame: Baseline and Post-Treatment (12 weeks)
Population: Completers
Measure: Number; unit: participants
Arm/Group | Placebo | QHS Zolpidem | Intermittant Zolpidem | CTRL
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 1 | 2 | 2 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | QHS Zolpidem | Intermittant Zolpidem | CTRL
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
About 25% of the target sample was obtained. As a result our capacity to detect trends and to calculate effect sizes was greatly diminished. Accordingly, our observations must be very limited in scope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No